CLINICAL TRIAL: NCT01107483
Title: Observe Change of Endotoxaemia and Related Mediators in Patients With Chronic HBV Infection
Brief Title: Observe Change of Endotoxaemia and Related Mediators in Patients With Chronic Hepatitis B Virus (HBV) Infection
Acronym: OCEHBV
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: The Third Affliated Hospital of Sun Yat-sen University, The Third Affliated Hospital of Sun Yat-sen University
Other Study IDs: endotoxaemiaobservation
Record Dates: First submitted 2010-04-16; First posted 2010-04-21 (Estimated); Last update posted 2010-05-07 (Estimated); Status verified 2010-01

CONDITIONS: Hepatitis B, Chronic
Keywords: endotoxaemia
MeSH Terms: conditions — Hepatitis B, Chronic; Endotoxemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- AC group: asymptomatic carriers
- CH group: patients with chronic hepatitis
- HC group: patients with hepatic cirrhosis
- ACLF group: patients with acute on chronic liver failure
- healthy control: healthy volunteers

SUMMARY:
This study was designed for changes in endotoxaemia, endotoxin-binding factors, sICAM-1 (soluble intracellular adhesion molecule-1), and cytokines during progression of chronic HBV infection. Patients with chronic HBV infection and healthy control are included. A limulus assay was used to measure plasma endotoxin level and ELISAs were used to measure the concentrations of interleukin-6 (IL-6), interleukin-10 (IL-10), tumor necrosis factor-α (TNFα), sICAM-1, and soluble CD14 (sCD14).

DETAILED DESCRIPTION:
1. Patients Patients with chronic HBV infection and healthy volunteers were enrolled. There were asymptomatic carriers group, patients with chronic hepatitis, patients with hepatic cirrhosis, and patients with acute on chronic liver failure.
2. Endotoxin assay Blood samples were obtained under aseptic conditions by peripheral venipuncture and using pyrogen-free syringes, needles, and glassware. Plasma samples were heated at 70℃ for 10 min. Plasma concentration was then measured in duplicate using a commercially available Limulus amebocyte lysate assay following the manufacturer's protocol.
3. ELISA ELISA kits were used to assess in duplicate the plasma concentrations of IL-6, IL-10, TNFα, sICAM-1 and sCD14.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HBV infection
* Diagnosis confirm to guideline of Chronic Hepatitis B and acute on chronic liver failure of the Asian Pacific Association for the Study of the Liver (APASL).

Exclusion Criteria:

* All the patients had no obvious mycotic infection, Gram-negative sepsis, or bacterial infection (except from the digestive system)
* Infection of hepatitis A, C, D, or E virus
* Autoimmune liver disease
* Alcoholic liver disease
* Metabolic liver disease
* Drug-induced liver injury
* Parasitic disease of the hepatobiliary system
* Malignancy
* Serious exacerbation of cardiovascular and respiratory system diseases

Ages: 24 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with chronic HBV infection admitted to The Third Affliated Hospital of Sun Yat-sen University
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2009-12; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
plasma levels of endotoxin | 4 months

SECONDARY OUTCOMES:
serum albumin level | 4 months
Plasma cytokine concentration | 4 months
  ELISA kits were used to assess in duplicate the plasma concentrations of IL-6, IL-10, TNFα, and sICAM-1 (Bender, Vienna, Austria).
serum low density lipoprotein (LDL) level | 4 months
serum high density lipoprotein (HDL) level | 4 months
plasma sCD14 level | 4 months
  ELISA kits were used to assess in duplicate the plasma concentrations of soluble CD14 (sCD14) (R&D Systems, Minneapolis, MN).

CONTACTS AND LOCATIONS:
Overall Officials: Gao Zhiliang, Professor, Study Chair — The Third Affliated Hospital of Sun Yat-sen University
Locations (1):
- The Third Affliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China